CLINICAL TRIAL: NCT03654287
Title: Exploring and Establishment of Multiple Organ Support Therapy（CELS）in Critically Ill Children
Brief Title: Exploring and Establishment of Combined Extracorporeal Life Support(CELS) in Critically Ill Children
Acronym: CELS
Status: Withdrawn | Type: Observational
Why Stopped: Interruption of financial support
Sponsor: Guoping Lu (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Guoping Lu, Director of pediatric Emergency and Critical Care Center. Children's Hospital Fudan University;Director of AHA Training Center for pediatric life support. Children's Hospital Fudan University, Children's Hospital of Fudan University
Organization: Children's Hospital of Fudan University (Other)
Other Study IDs: fdpicu-02
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Sepsis; Critical Illness; MODS
Keywords: sepsis; CRRT; ECMO; CELS
MeSH Terms: conditions — Sepsis; Critical Illness; Multiple Organ Failure | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Treatment with CPFA: The critically ill children who treated by CRRT and CRRT mode is decide as CPFA.
  Interventions: Other: Treatment
- Treatment with TPE+CVVHDF: The critically ill children who treated by CRRT and CRRT mode is decide as TPE+CVVHDF.
  Interventions: Other: Treatment
- Treatment with CVVHDF: The critically ill children who treated by CRRT and CRRT mode is decide as CVVHDF.
  Interventions: Other: Treatment
- Treatment without CRRT/ECMO: The critically ill children who are not treated by CRRT or ECMO.
- Treatment with ECMO: The critically ill children who are treated by ECMO whether treated by CRRT
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — The CELS way to intervene severe sepsis and refractory shock
  Groups: Treatment with CPFA; Treatment with CVVHDF; Treatment with ECMO; Treatment with TPE+CVVHDF

SUMMARY:
Multiple organ failure (MODS) is still the leading cause of death in children in ICU. The treatment of MODS is mainly organ function monitoring and organ replacement therapy. Life support technology in vitro mainly includes mechanical ventilation, continuous renal replacement therapy (CRRT), non-biological artificial liver and extracorporeal membrane oxygenation technology (ECMO). However, critically ill patients who have multiple organ failure often require multiple organ support meanwhile. Combined extracorporeal life support (CELS) is still in its infancy to be applied in the treatment of critical illness due to nonstandard technology and theory without key breakthroughs and evidence-based medicine in the treatment of severe children organ failure.Solving the system problems supported by CELS can effectively reduce the mortality and disability rate of critically ill children and enhance health care in Shanghai, even across China.

DETAILED DESCRIPTION:
The whole study is described below. To investigate the timing ,curative effect and mode of CRRT and ECMO treatment for critically ill children,we choose sepsis children especially those who are combined with septic shock as research object.

Furthermore,refractory shock is the therapeutic indications of ECMO. According to their clinical manifestation and severity of the disease,they are treated by CRRT or/with ECMO in a non-randomized way.

Comparing the laboratory index and prognosis of critically ill children treated by CRRT and those treated by ECMO,we aim to investigate the the timing ,curative effect of ECMO in the treatment of septic shock especially refractory shock.

The critically ill children who treated by CRRT are divided into three groups according to their treatment mode of CRRT. The laboratory index and prognosis are also be compared to investigate curative effect of CRRT in the treatment of septic shock.

The study also include severe sepsis children without CRRT or ECMO treatment as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Children with severe sepsis and refractory shock admitted to the PICU of four study centers.

The informed consent of the guardians

Exclusion Criteria:

* active hemorrhage difficult catheter placing Irreversible brain damage patients enrolled in other clinic trial

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with severe sepsis and refractory shock admitted to the PICU of four study centers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
survival rate | 28 days
  The survival rate of children in 28 days after their hospital discharged.

SECONDARY OUTCOMES:
Pediatric Risk of Mortality score （PRISM III） | the first 24 hours after admitted to PICU
  The PRISM score is a quantification of physiologic status using predetermined physiologic variables and their ranges that use categorical variables to facilitate accurate estimation of mortality risk.The PRISM components were separated into cardiovascular (heart rate, systolic blood pressure, and temperature), neurologic ( pupillary reactivity and mental status), respiratory (arterial Po2, pH, Pco2, and total bicarbonate), chemical (glucose, potassium, blood urea nitrogen, and creatinine), and hematologic (WBC count, platelet count, prothrombin, and partial thromboplastin time) component.The score above 10 indicates a poor prognosis and higher mortality of critical ill children. The score below 10 indicates a relatively favorable prognosis and lower mortality .
ECMO weaning rate | 48 hours
  The success of ECMO weaning is defined as the survival of patients after ECMO is wean for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guoping LU, doctor, Principal Investigator — Children's Hospital of Fundan University
Locations (1):
- Children'S Hosptial of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided